CLINICAL TRIAL: NCT05020782
Title: Open-label, Prospective, Phase II Descriptive Pilot Trial of Belimumab Therapy for Refractory and/or Non-criteria Manifestations of Antiphospholipid Syndrome
Brief Title: The BeLimumab Antiphospholipid Syndrome Trial (BLAST)
Acronym: BLAST
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Turin, Italy (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APSGB01
Record Dates: First submitted 2021-07-29; First posted 2021-08-25 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2022-05

CONDITIONS: Antiphospholipid Syndrome
MeSH Terms: conditions — Antiphospholipid Syndrome | interventions — belimumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention Arm (Experimental): INTERVENTION DRUG: BELIMUMAB 10 MG/KG
  Interventions: Drug: Belimumab

INTERVENTIONS:
Drug: Belimumab — INTERVENTION DRUG: BELIMUMAB 10 MG/KG

SUMMARY:
AIM: The primary objective of the BeLimumab Antiphospholipid Syndrome Trial (BLAST) is to evaluate the safety and tolerability of belimumab for up to 24 months in patients with persistent aPL positivity and clinical features attributable to aPL that are resistant to warfarin and/or heparin.

ELIGIBILITY:
Inclusion Criteria:

• Positive aPL profile defined as: Positive lupus anticoagulant test as defined by the International Society on Thrombosis and Haemostasis, on two or more occasions, at least 12 weeks apart and/or Positive anticardiolipin antibody (aCL) immunoglobulin G(Ig)G/M/A isotype, present in > 40U, on two or more occasions, at least 12 weeks apart and/or Positive anti-β2-glycoprotein-I (aβ2GPI) IgG/M/A isotype, present in > 40U, on two or more occasions, at least 12 weeks apart

AND

• Clinical features attributable to aPL that are resistant to warfarin and/or heparin:

* Recurrent thrombosis despite ongoing anticoagulation and/or
* Persistent thrombocytopenia and/or
* Persistent autoimmune hemolytic anemia and/or
* Cardiac valve disease and/or
* Chronic skin ulcers and/or
* Renal thrombotic microangiopathy and/or
* Cognitive dysfunction with/without white matter changes

Exclusion Criteria:

* >=4/11 American College of Rheumatology Classification Criteria for SLE
* Acute thrombosis (arterial or venous acute thrombosis diagnosis less than 30 days before study screening)
* History of stroke Acute or chronic pancreatitis
* Pregnancy
* Have a history of malignant neoplasm within the last 5 years except basal cell or squamous cell carcinoma of the skin treated with local resection only or carcinoma in situ of the uterine cervix treated locally and with no evidence of metastatic disease for 3 years
* Have evidence of serious suicide risk including any history of suicidal behaviour in the last 6 months and/or any suicidal ideation in the last 2 months or who in the investigator's judgment, poses a significant suicide risk
* Have a history of a primary immunodeficiency
* Have a significant IgG deficiency (IgG level < 400 mg/dL)
* Have an IgA deficiency (IgA level < 10 mg/dL)
* Known active bacterial, viral fungal mycobacterial, or other infection
* Infection history:
* Currently on any suppressive therapy for a chronic infection (such as tuberculosis, pneumocystis, cytomegalovirus, herpes simplex virus, herpes zoster and atypical mycobacteria)
* Hospitalization for treatment of infection within 60 days of Day 0.
* Use of parenteral (IV or IM) antibiotics (anti-bacterial, antiviral, anti-fungal, or antiparasitic agents) within 60 days of Day 0
* Have current drug or alcohol abuse or dependence, or a history of drug or alcohol abuse or dependence within 365 days prior to Day 0
* Have a historically positive HIV test or test positive at screening for HIV
* Hepatitis status:
* Serologic evidence of current or past Hepatitis B (HB) infection based on the results of testing for HBsAg and HBcAb as follows:
* Patients positive for HBsAg or HBcAb are excluded
* Positive test for Hepatitis C antibody
* Have a history of an anaphylactic reaction to parenteral administration of contrast agents, human or murine proteins or monoclonal antibodies
* Have any other clinically significant abnormal laboratory value in the opinion of the investigator
* If Women of Child-Bearing Potential (WCBP) are included, please see special instructions below.
* Have any intercurrent significant medical or psychiatric illness that the investigator considers would make the candidate unsuitable for the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Adverse Events | 104 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
The Efficacy of Belimumab-thrombocytopenia | 104 weeks
  Outcome measures scored as complete response (CR), partial (PR), and none (NR) at 24, 52, 104 weeks. For thrombocytopenia, CR defined as a platelet count of ≥150×109/μl,PR as 100-149,and NR as <100.
The Efficacy of Belimumab-CVD | 104 weeks
  Outcome measures scored as complete response (CR), partial (PR), and none (NR) at 24, 52, 104 weeks.For CVD,CR defined as the disappearance of cardiac lesions, PR as 50%improvement,and NR as no change.
The Efficacy of Belimumab-renal involvement | 104 weeks
  Outcome measures scored as complete response (CR), partial (PR), and none (NR) at 24, 52, 104 weeks. For aPL nephropathy, CR defined as a normal serum creatinine level, inactive urinary sediment, and urinary protein: creatinine 0.5;PR as a serum cr level 15% above baseline, RBCs per high-power field 50% above baseline with no casts, 50%improvement in the urinary prt:cr, and estimated GFR 10%above baseline; and NR as the absence of C/PR.
The Efficacy of Belimumab-cognitive impairment | 104 weeks
  Outcome measures scored as complete response (CR), partial (PR), and none (NR) at 24, 52, 104 weeks. For cognitive dysfunction,CR defined as normalization of the cognitive impairment index with 50%improvement,PR as abnormal index with 50%, and NR as no change.
The Efficacy of Belimumab-thrombosis | 104 weeks
  Rate of documented thrombotic events
Change in aPL profile | 104 weeks
  Change in aPL levels at 24, 52, 104 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- San Giovanni Bosco Hospital, Turin, Piedmont, Italy